CLINICAL TRIAL: NCT04824482
Title: GAIT Recovery in Patients aFter Acute Ischemic STroke: A Randomized Comparison of Robot-assisted and Therapist-assisted Gait Training on a Treadmill.
Brief Title: Gait Recovery in Patients After Acute Ischemic Stroke
Acronym: GAITFAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Barbora Kolarova, Head of Kinesiology Laboratory, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NU21-04-00375
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Stroke rehabilitation; Physical Therapy; Gait; Exoskeleton Device; Walking speed; Gait Analysis; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: All participants will be randomly assigned to two parallel intervention groups for the duration of study. Thirty patients from each intervention group will be randomized to multimodal MRI of brain.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted treadmill gait training (RTGT) (Experimental): Locomotor training guided by the robotic device (Lokomat Hocoma) according to a pre-programmed gait pattern with the help of robot-driven exoskeleton orthoses. The process of gait training is automated and controlled by a computer under supervision of a physiotherapist.
  Interventions: Other: Robot-assisted treadmill gait training (RTGT)
- Therapist-assisted treadmill gait training (TTGT) (Active Comparator): Locomotor training via a repetitive execution of walking movements manually guided by a physiotherapist during treadmill gait training.
  Interventions: Other: Therapist-assisted treadmill gait training (TTGT)

INTERVENTIONS:
Other: Robot-assisted treadmill gait training (RTGT) — Locomotor training guided by the robotic device (Lokomat Hocoma) according to a pre-programmed gait pattern with the help of robot-driven exoskeleton orthoses. The process of gait training is automated and controlled by a computer under supervision of a physiotherapist.
  Arms: Robot-assisted treadmill gait training (RTGT)
Other: Therapist-assisted treadmill gait training (TTGT) — Locomotor training via a repetitive execution of walking movements manually guided by a physiotherapist during treadmill gait training.
  Arms: Therapist-assisted treadmill gait training (TTGT)

SUMMARY:
More than 80% of ischemic stroke (IS) patients have some walking disability, which restricts their independence in the activities of daily living. Physical therapy (PT) significantly contributes to gait recovery in patients after IS. However, it remains unclear, what type of gait training is more effective and which factors may have impact on gait recovery. Two hundred fifty IS patients will be enrolled to undergo a 2-week intensive inpatient rehabilitation including randomly assigned robot-assisted treadmill gait training (RTGT) or therapist-assisted treadmill gait training (TTGT). A detailed clinical and laboratory assessment of gait quality, as well as the degree of neurological impairment, quality of life, cognition and depression will be performed in all patients during the study. We hypothesize that these variables may also affect gait recovery in patients after IS. In a randomly selected 60 enrolled patients, a multi-modal magnetic resonance imaging (MRI), including functional MRI, will be performed to assess neural correlates and additional predictors of gait recovery.

DETAILED DESCRIPTION:
One hundred twenty consecutive first ever ischemic stroke patients classified as dependent walkers (Functional Ambulatory Category interval <1,3>) will be enrolled in the randomized blinded single center prospective clinical trial GAITFAST with a randomization either for robot-assisted treadmill gait training (RGT) or therapist-assisted treadmill gait training (TTGT) after acute phase (5-10 days after stroke onset). All enrolled patients will undergo a 2-week intensive inpatient rehabilitation including randomly assigned TTGT or RTGT followed with clinical visits (at the beginning of inpatient rehabilitation, at discharge, and three and six months after enrollment in the study). Each clinical visit will include detailed clinical functional assessments, assessment of spatiotemporal and kinetic gait parameters, assessment of neurological impairment, assessment of quality of life, cognition and depression. In 60 randomly selected enrolled IS patients, a repeated multi-modal magnetic resonance imaging (MRI) including functional MRI (fMRI) will be performed during the study follow-up to identify brain structures with possible impact on gait recovery.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke detected on magnetic resonance imaging (MRI) with NIHSS score 1-12 points at the time of enrolment
* Lower limb movement impairment with a score of at least 1 point on the NIH Stroke Scale (NIHSS) at the time of enrolment
* Dependency in walking according to Functional Ambulatory Category (FAC) with score interval <1,3> (supervision or assistance, or both, must be given in performing walking)

Exclusion Criteria:

* Previous history of any stroke, either ischemic or hemorrhagic
* Other diseases modifying or limiting walking ability, currently receiving rehabilitation or participation in another study
* Significant/symptomatic ischemic heart disease or significant/symptomatic peripheral arterial disease
* Obesity (BMI ≥ 40), or weight higher than 110 kg (weight limit for the robot-assisted gait training)
* Sensory aphasia with the inability to understand having been verified by a certified speech therapist.
* Moderate or severe depression present at the time of enrolment assessed using the Beck scale, with a score above 10.
* Known cognitive impairment
* Previous disability or dependence in the daily activities assessed using the modified Rankin Scale with a score of 3 and more points
* Currently receiving dialysis
* Diagnosed and/or receiving treatment for cancer
* Presence of other orthopedic or neurological conditions affecting the lower extremities
* For fMRI: Pregnancy; electronic implants, including cochlear implant, pacemaker, neurostimulator; incompatible metallic implants, including aneurysm clip; metallic intraocular foreign body; large tattoos; unremovable piercing; body weight over 150 kg; known claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in gait speed during overground walking | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Gait speed will be measured using the 10 Meters Walking Test (performance measure used to assess walking speed in meters per second over a short distance). The subject will be asked to walk for a distance of 10 meters at his/her comfortable speed. The time will be measured for the distance of the middle six meters, which will allow walk acceleration and deceleration. Each patient will perform two trials with a calculation of mean time value. If physical assistance of another person (to prevent a fall or collapsing) is needed for a patient to complete the test, the level of assistance provided will be documented. Usage of any assistive device and/or bracing (that patients are currently using for walking and are needed to complete the test) will be also documented.

SECONDARY OUTCOMES:
Change in National Institute of Health Stroke Scale (NIHSS) | Enrollment, baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  NIHSS is used to objectively quantify the impairment caused by a stroke.
Change in gait speed (km/h) during patients´ comfort speed | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Gait speed will be assessed by instrumented treadmill gait analysis system (Zebris Medical GmbH, FDM-T system).
Change in gait cadence (steps/min) during patients´ comfort speed | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Gait cadence will be assessed by instrumented treadmill gait analysis system (Zebris Medical GmbH, FDM-T system).
Change in paretic and non-paretic leg step length (cm) during patients´ comfort speed | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Change in paretic and non-paretic leg step length will be assessed by instrumented treadmill gait analysis system (Zebris Medical GmbH, FDM-T system).
Change in duration of stance phase as percentage of gait cycle (%) for paretic and non-paretic limb during patients´ comfort speed | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Change in duration of stance phase will be assessed by instrumented treadmill gait analysis system (Zebris Medical GmbH, FDM-T system).
Change in double stance phase as percentage of gait cycle (%) during patients´ comfort speed | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Change in double stance phase will be assessed by treadmill gait analysis system (Zebris Medical GmbH, FDM-T system).
Change in ground reaction force (N) for paretic and non-paretic limb during patients' comfort speed | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Change in ground reaction force will be assessed by instrumented treadmill gait analysis system (Zebris Medical GmbH, FDM-T system).
Change in plantar pressure distribution (N/cm2) for paretic and non-paretic limb during patients´ comfort speed | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Change in plantar pressure distribution will be assessed by instrumented treadmill gait analysis system (Zebris Medical GmbH, FDM-T system).
Change in Functional Ambulatory Category FAC | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Functional walking test that assess gait ability with 6 levels ranging from 0 to 5 on the basis of the amount of physical support required.
Change in Fugl-Meyer Assessment | baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Fugl-Meyer Assessment uses to examine the sensory-motor function and coordination of affected lower extremity.
Change in functional magnetic resonance imaging activation magnitude | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Functional MRI activation magnitude, calculated as difference in BOLD signal between task and rest, will be assessed within pre-defined gait-related brain regions of interest (ROIs), i.e., sensorimotor cortex, premotor cortex, supplementary motor area, brainstem and cerebellum. Change in these ROI parameters over time will be statistically tested within group and the regional post-training minus pre-training difference in each group will be submitted to between-group analysis.
Change in functional magnetic resonance imaging activation volume | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Functional MRI activation volume, summed over significantly activated voxels, will be assessed within pre-defined gait-related brain regions of interest (ROIs), i.e., sensorimotor cortex, premotor cortex, supplementary motor area, brainstem and cerebellum. Change in these ROI parameters over time will be statistically tested within group and the regional post-training minus pre-training difference in each group will be submitted to between-group analysis.

OTHER OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) Test | Enrollment, baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  MoCA is cognitive screening test designed to detection cognitive impairment. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation.
Change in Modified Rankin Scale | Enrollment, baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Scale used for measuring the degree of disability or dependence in the daily activities in patients after stroke. Most widely used clinical outcome measure after stroke. Scale has six points and higher score means worse outcome; minimum is 0 points indicating no symptoms at all and maximum is 6 points indicating death.
Change in Barthel index | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Barthel index is scale used to measure performance in activities of daily living (ADL). The maximum score is 100 points.
Change in Timed Up and Go test | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Clinical test used to assess a person's mobility which requires both static and dynamic balance. The objective of this test is to determine fall risk and measure the progress of balance, sit to stand and walking.
Change in Lower limb muscle strength assessment | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Medical Research Council Scale for Muscle Strength will be used for assessment
Change in lower limb muscles activity (medial gastrocnemius, tibialis anterior, quadriceps, hamstrings) during the 10 Meter Walk | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Change in lower limb muscles activity (medial gastrocnemius, tibialis anterior, quadriceps, hamstrings) will be assessed by surface electromyography (Delsys Trigno EMG/IMU sensors).
Change in lower limb muscles activity (medial gastrocnemius, tibialis anterior, quadriceps, hamstrings) during treadmill gait | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Change in lower limb muscles activity (medial gastrocnemius, tibialis anterior, quadriceps, hamstrings) will be assessed by surface electromyography (Delsys Trigno EMG/IMU sensors).
Change in Beck Depression Inventory Scale | Enrollment, after three weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  A 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Each item (question) had a set of at least four possible responses, ranging in intensity. 0-9: indicates minimal depression and 30-63 points indicates severe depression. Higher total scores indicate more severe depressive symptoms.
Change in EQ-5D-3L Questionnaire | Baseline (before beginning of inpatient RHB), after two weeks (at the end of inpatient RHB), and in follow-up (after three and six months after stroke onset)
  Standard layout for recording an adult person's current self-reported health state. Consists of a standard format for respondents to record their health state according to the EQ-5D-3L descriptive system and the EQ VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Hlustik, MD, PhD, Study Chair — Palacky University
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

REFERENCES:
- [Background] Norrving B, Kissela B. The global burden of stroke and need for a continuum of care. Neurology. 2013 Jan 15;80(3 Suppl 2):S5-12. doi: 10.1212/WNL.0b013e3182762397. PMID 23319486
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Gordon NF, Gulanick M, Costa F, Fletcher G, Franklin BA, Roth EJ, Shephard T; American Heart Association Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Physical activity and exercise recommendations for stroke survivors: an American Heart Association scientific statement from the Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Circulation. 2004 Apr 27;109(16):2031-41. doi: 10.1161/01.CIR.0000126280.65777.A4. No abstract available. PMID 15117863
- [Background] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK; LEAPS Investigative Team. Protocol for the Locomotor Experience Applied Post-stroke (LEAPS) trial: a randomized controlled trial. BMC Neurol. 2007 Nov 8;7:39. doi: 10.1186/1471-2377-7-39. PMID 17996052
- [Background] Alia C, Spalletti C, Lai S, Panarese A, Lamola G, Bertolucci F, Vallone F, Di Garbo A, Chisari C, Micera S, Caleo M. Neuroplastic Changes Following Brain Ischemia and their Contribution to Stroke Recovery: Novel Approaches in Neurorehabilitation. Front Cell Neurosci. 2017 Mar 16;11:76. doi: 10.3389/fncel.2017.00076. eCollection 2017. PMID 28360842
- [Background] Nudo RJ. Recovery after brain injury: mechanisms and principles. Front Hum Neurosci. 2013 Dec 24;7:887. doi: 10.3389/fnhum.2013.00887. PMID 24399951
- [Background] Kwakkel G, Kollen B, Lindeman E. Understanding the pattern of functional recovery after stroke: facts and theories. Restor Neurol Neurosci. 2004;22(3-5):281-99. PMID 15502272
- [Background] Pollock A, Farmer SE, Brady MC, Langhorne P, Mead GE, Mehrholz J, van Wijck F. Interventions for improving upper limb function after stroke. Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD010820. doi: 10.1002/14651858.CD010820.pub2. PMID 25387001
- [Background] Kerr AL, Cheng SY, Jones TA. Experience-dependent neural plasticity in the adult damaged brain. J Commun Disord. 2011 Sep-Oct;44(5):538-48. doi: 10.1016/j.jcomdis.2011.04.011. Epub 2011 May 6. PMID 21620413
- [Background] Kleim JA, Barbay S, Nudo RJ. Functional reorganization of the rat motor cortex following motor skill learning. J Neurophysiol. 1998 Dec;80(6):3321-5. doi: 10.1152/jn.1998.80.6.3321. PMID 9862925
- [Background] Wallard L, Dietrich G, Kerlirzin Y, Bredin J. Effects of robotic gait rehabilitation on biomechanical parameters in the chronic hemiplegic patients. Neurophysiol Clin. 2015 Sep;45(3):215-9. doi: 10.1016/j.neucli.2015.03.002. Epub 2015 Sep 14. PMID 26381192
- [Background] Luft AR, Macko RF, Forrester LW, Villagra F, Ivey F, Sorkin JD, Whitall J, McCombe-Waller S, Katzel L, Goldberg AP, Hanley DF. Treadmill exercise activates subcortical neural networks and improves walking after stroke: a randomized controlled trial. Stroke. 2008 Dec;39(12):3341-50. doi: 10.1161/STROKEAHA.108.527531. Epub 2008 Aug 28. PMID 18757284
- [Background] Enzinger C, Dawes H, Johansen-Berg H, Wade D, Bogdanovic M, Collett J, Guy C, Kischka U, Ropele S, Fazekas F, Matthews PM. Brain activity changes associated with treadmill training after stroke. Stroke. 2009 Jul;40(7):2460-7. doi: 10.1161/STROKEAHA.109.550053. Epub 2009 May 21. PMID 19461018
- [Background] Burke E, Dobkin BH, Noser EA, Enney LA, Cramer SC. Predictors and biomarkers of treatment gains in a clinical stroke trial targeting the lower extremity. Stroke. 2014 Aug;45(8):2379-84. doi: 10.1161/STROKEAHA.114.005436. Epub 2014 Jun 24. PMID 25070961
- [Background] Jahn K, Deutschlander A, Stephan T, Strupp M, Wiesmann M, Brandt T. Brain activation patterns during imagined stance and locomotion in functional magnetic resonance imaging. Neuroimage. 2004 Aug;22(4):1722-31. doi: 10.1016/j.neuroimage.2004.05.017. PMID 15275928
- [Background] Maidan I, Rosenberg-Katz K, Jacob Y, Giladi N, Hausdorff JM, Mirelman A. Disparate effects of training on brain activation in Parkinson disease. Neurology. 2017 Oct 24;89(17):1804-1810. doi: 10.1212/WNL.0000000000004576. Epub 2017 Sep 27. PMID 28954877
- [Background] Leonard G, Lapierre Y, Chen JK, Wardini R, Crane J, Ptito A. Noninvasive tongue stimulation combined with intensive cognitive and physical rehabilitation induces neuroplastic changes in patients with multiple sclerosis: A multimodal neuroimaging study. Mult Scler J Exp Transl Clin. 2017 Feb 1;3(1):2055217317690561. doi: 10.1177/2055217317690561. eCollection 2017 Jan-Mar. PMID 28607750
- [Background] Sacheli LM, Zapparoli L, Preti M, De Santis C, Pelosi C, Ursino N, Zerbi A, Stucovitz E, Banfi G, Paulesu E. A functional limitation to the lower limbs affects the neural bases of motor imagery of gait. Neuroimage Clin. 2018 Jul 5;20:177-187. doi: 10.1016/j.nicl.2018.07.003. eCollection 2018. PMID 30094167
- [Background] la Fougere C, Zwergal A, Rominger A, Forster S, Fesl G, Dieterich M, Brandt T, Strupp M, Bartenstein P, Jahn K. Real versus imagined locomotion: a [18F]-FDG PET-fMRI comparison. Neuroimage. 2010 May 1;50(4):1589-98. doi: 10.1016/j.neuroimage.2009.12.060. Epub 2009 Dec 23. PMID 20034578
- [Background] Mehrholz J, Thomas S, Werner C, Kugler J, Pohl M, Elsner B. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2017 May 10;5(5):CD006185. doi: 10.1002/14651858.CD006185.pub4. PMID 28488268
- [Background] Kim HY, Shin JH, Yang SP, Shin MA, Lee SH. Robot-assisted gait training for balance and lower extremity function in patients with infratentorial stroke: a single-blinded randomized controlled trial. J Neuroeng Rehabil. 2019 Jul 29;16(1):99. doi: 10.1186/s12984-019-0553-5. PMID 31358017
- [Background] Moucheboeuf G, Griffier R, Gasq D, Glize B, Bouyer L, Dehail P, Cassoudesalle H. Effects of robotic gait training after stroke: A meta-analysis. Ann Phys Rehabil Med. 2020 Nov;63(6):518-534. doi: 10.1016/j.rehab.2020.02.008. Epub 2020 Mar 27. PMID 32229177
- [Background] Kahn LE, Lum PS, Rymer WZ, Reinkensmeyer DJ. Robot-assisted movement training for the stroke-impaired arm: Does it matter what the robot does? J Rehabil Res Dev. 2006 Aug-Sep;43(5):619-30. doi: 10.1682/jrrd.2005.03.0056. PMID 17123203
- [Background] Smith MC, Barber PA, Stinear CM. The TWIST Algorithm Predicts Time to Walking Independently After Stroke. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):955-964. doi: 10.1177/1545968317736820. Epub 2017 Nov 1. PMID 29090654
- [Background] Middleton A, Fritz SL, Lusardi M. Walking speed: the functional vital sign. J Aging Phys Act. 2015 Apr;23(2):314-22. doi: 10.1123/japa.2013-0236. Epub 2014 May 2. PMID 24812254
- [Background] Richards JD, Pramanik A, Sykes L, Pomeroy VM. A comparison of knee kinematic characteristics of stroke patients and age-matched healthy volunteers. Clin Rehabil. 2003 Aug;17(5):565-71. doi: 10.1191/0269215503cr651oa. PMID 12952165
- [Background] Jahn K, Deutschlander A, Stephan T, Kalla R, Wiesmann M, Strupp M, Brandt T. Imaging human supraspinal locomotor centers in brainstem and cerebellum. Neuroimage. 2008 Jan 15;39(2):786-92. doi: 10.1016/j.neuroimage.2007.09.047. Epub 2007 Oct 10. PMID 18029199
- [Background] Hok P, Opavsky J, Labounek R, Kutin M, Slachtova M, Tudos Z, Kanovsky P, Hlustik P. Differential Effects of Sustained Manual Pressure Stimulation According to Site of Action. Front Neurosci. 2019 Jul 17;13:722. doi: 10.3389/fnins.2019.00722. eCollection 2019. PMID 31379481
- [Background] Schwartz I, Sajin A, Fisher I, Neeb M, Shochina M, Katz-Leurer M, Meiner Z. The effectiveness of locomotor therapy using robotic-assisted gait training in subacute stroke patients: a randomized controlled trial. PM R. 2009 Jun;1(6):516-23. doi: 10.1016/j.pmrj.2009.03.009. PMID 19627940
- [Background] Tilson JK, Sullivan KJ, Cen SY, Rose DK, Koradia CH, Azen SP, Duncan PW; Locomotor Experience Applied Post Stroke (LEAPS) Investigative Team. Meaningful gait speed improvement during the first 60 days poststroke: minimal clinically important difference. Phys Ther. 2010 Feb;90(2):196-208. doi: 10.2522/ptj.20090079. Epub 2009 Dec 18. PMID 20022995
- [Background] Holden MK, Gill KM, Magliozzi MR. Gait assessment for neurologically impaired patients. Standards for outcome assessment. Phys Ther. 1986 Oct;66(10):1530-9. doi: 10.1093/ptj/66.10.1530. PMID 3763704
- [Derived] Kolarova B, Sanak D, Hlustik P, Kolar P. Randomized Controlled Trial of Robot-Assisted Gait Training versus Therapist-Assisted Treadmill Gait Training as Add-on Therapy in Early Subacute Stroke Patients: The GAITFAST Study Protocol. Brain Sci. 2022 Dec 3;12(12):1661. doi: 10.3390/brainsci12121661. PMID 36552120